CLINICAL TRIAL: NCT07209852
Title: Safety, Performance, and Clinical Benefit of Pacing the Left Bundle Branch Area - Post-Market Clinical Follow-up (SEPTA PMCF)
Brief Title: Safety, Performance, and Clinical Benefit of Pacing the Left Bundle Branch Area - Post-Market Clinical Follow-up
Acronym: SEPTA PMCF
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: SEPTA PMCF - C2211
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bradycardia; Atrioventricular Block; Sinus Node Dysfunction; Bundle-Branch Block
Keywords: Left Bundle Branch Area Pacing (LBBAP); INGEVITY+ Lead; Pacemaker; Cardiac Pacing; Conduction System Pacing; Ventricular Synchrony; Post-Market Clinical Follow-up
MeSH Terms: conditions — Bradycardia; Atrioventricular Block; Sick Sinus Syndrome; Bundle-Branch Block | interventions — Device Lead Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients receiving INGEVITY+ lead for left bundle branch area pacing: This group includes adult patients with bradycardia who are indicated for a Boston Scientific pacemaker system. All participants will undergo implantation of an INGEVITY+ pace/sense lead in the left bundle branch area (LBBAP) with a compatible Boston Scientific pacemaker.
  Interventions: Device: Pacemaker lead

INTERVENTIONS:
Device: Pacemaker lead — The pacemaker lead under investigation is a bipolar, steroid-releasing pacemaker electrode with active fixation (IS-1 connection) designed for chronic stimulation and sensing in the right atrium, right ventricle or left bundle branch area (LBBA). In this study, the lead is implanted in the LBBA and connected to a single- or dual-chamber pacemaker. Implantation is performed using a compatible, CE-marked catheter for pacemaker implantation.
  Other Names: Bradycardia pacemaker system; Left Bundle Branch Area Pacing (LBBAP) Lead

SUMMARY:
The goal of this observational post-market clinical Follow-up study is to learn about the long-term safety, performance, and clinical benefits of pacing the left bundle branch area (LBBAP) using the INGEVITY+ pacemaker lead in patients with bradycardia who need a pacemaker.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects intended to undergo initial (de novo) pacing system implant using the INGEVITY+ lead in the left bundle branch area (LBBA) and a Boston Scientific single or dual- chamber pacemaker (Note: no prior attempted pacing system components);
2. Subjects who are indicated for and will receive a Boston Scientific pacemaker system (including the single or dual chamber pacemaker and an INGEVITY+ lead in the LBBA location) for one of the following medical conditions:

   1. Symptomatic paroxysmal or permanent second- or third-degree AV block,
   2. Symptomatic bilateral bundle branch block,
   3. Symptomatic paroxysmal or transient sinus node dysfunction with or without associated AV conduction disorders (i.e., sinus bradycardia, sinus arrest, sinoatrial [SA] block),
   4. Bradycardia-tachycardia syndrome, to prevent symptomatic bradycardia or some forms of symptomatic tachyarrhythmias,
   5. Neurovascular (vasovagal) syndromes or hypersensitive carotid sinus syndromes,
   6. Adaptive-rate pacing for patients exhibiting chronotropic incompetence and who may benefit from increased pacing rates concurrent with increases in minute ventilation and/or level of physical activity.

      Dual-chamber and atrial tracking modes are also indicated for patients who may benefit from maintenance of AV synchrony. Dual chamber modes are specifically indicated for treatment of the following:
   7. Conduction disorders that require restoration of AV synchrony, including varying degrees of AV block,
   8. VVI intolerance (i.e., pacemaker syndrome) in the presence of persistent sinus rhythm,
   9. Low cardiac output or congestive heart failure secondary to bradycardia;
3. Subjects willing and capable of providing informed consent and participating in all testing and clinic visits associated with the clinical study at an approved clinical study location and at the intervals defined by protocol;
4. Subjects who are ≥18 years of age, and of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects meeting guideline indications for cardiac resynchronization therapy (CRT) in the absence of a bradycardia indication;
2. Subjects with a known or suspected sensitivity to dexamethasone acetate (DXA);
3. Subjects with a Mechanical Tricuspid Valve;
4. Subjects requiring hemodialysis or peritoneal dialysis;
5. Subject has or has had implanted any pacemaker, ICD system, including subcutaneous, transvenous or leadless systems (Note: except for temporary pacing wire at time of enrollment) or CRT system;
6. Subjects currently on an active organ transplant list;
7. Subject referred to or admitted for hospice care;
8. Subjects with a documented life expectancy of less than 12 months;
9. Subjects enrolled in any other concurrent study (unless prior approval is received from the Sponsor);
10. Subjects who are, or plan to become pregnant during the course of the study or are breastfeeding at time of enrollment;
11. Subjects who are unable or unwilling to comply with the follow-up schedule, including those living at such a distance from the investigational site that attending follow-up visits would be unusually difficult or burdensome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in SEPTA PMCF will be selected from the physician investigator's general patient population with a brady pacing indication for single or dual-chamber pacemaker implantation where LBBAP is preferred. Diverse racial and gender patient consideration should be implemented when determining potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
LBBA Implant Success Rate | At the time of implant procedure (Day 0).
  Percentage of subjects in whom the INGEVITY+ lead is successfully implanted in the left bundle branch area (LBBA). Implant success is determined by ECG and procedural criteria, as defined per protocol.
Maintenance of Ventricular Synchrony (Paced QRS Duration) | From implant through 3-year follow-up.
  Mean paced QRS duration measured by 12-lead ECG to assess preservation of ventricular synchrony.

OTHER OUTCOMES:
Lead-related Complication-Free Rate | From implant through 3 years.
  Freedom from lead-related complications (death, serious injury, invasive correction, or permanent loss of device function).

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Wauters, MD, PhD, Principal Investigator — Clinique St-Pierre Ottignies
Locations (13):
- Belgium (2):
  - St. Jan-Hospital, Bruges
  - Clinique Saint-Pierre Ottignies-Hospital, Brussels
- France (2):
  - CHRU de Lille, Lille
  - Hospital Europeen Georges-Pompidou (HEGP), Paris
- Germany (2):
  - Marienhospital-Hospital, Osnabrück, Lower Saxony
  - Saarland University Hospital, Homburg, Saarland
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Ferrara-Hospital, Ferrara, Emilia-Romagna
  - Azienda Ospedaliera Ospedale Niguarda Ca Granda, Milan
  - AOU Maggiore, Novara
- Spain (2):
  - Virgen de las Nieves University Hospital, Granada
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Inselspital Bern, Bern, Switzerland
- East Surrey Hospital, Redhill, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No